CLINICAL TRIAL: NCT05395962
Title: Electrochemotherapy With Carboplatinum Plus Bleomycin Versus Bleomycin Alone in Vulvar Cancer: the ElechtraPlatinum Study. A Randomized Controlled Trial
Brief Title: Electrochemotherapy With Carboplatinum Plus Bleomycin Versus Bleomycin Alone in Vulvar Cancer
Acronym: Elechtra
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Anna Myriam Perrone, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41/2022/Farm/AOUBo
Record Dates: First submitted 2022-05-11; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Vulvar Cancer
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Carboplatin; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLM (Active Comparator)
  Interventions: Drug: Bleomycin
- BLM+CBP (Experimental)
  Interventions: Drug: Carboplatin; Drug: Bleomycin

INTERVENTIONS:
Drug: Carboplatin — treatment with bleomycin and carboplatin in association with electroporation
  Arms: BLM+CBP
Drug: Bleomycin — treatment with bleomycin in association with electroporation

SUMMARY:
Patients with vulvar cancer who underwent multiple treatments (surgery and radiation therapy or chemoradiation, radiation therapy or chemoradiation and chemotherapy), or patients not eligible for standard therapies.

The study aims to:

* Evaluate the oncology response to electroporation after administration of Bleomycin (BLM) + carboplatinum (CBP )to BLM alone in terms of local progression-free survival (LPFS) in women with relapsed vulvar cancer after multimodal treatments.
* Compare quality of life (HR-QoL) in the two groups of patients with questionnaires (FACT-V, FACT-PAL, E5-5L-D5).
* To compare Overall Survival in the two study arms.
* To compare local and systemic toxicity, morbidity and mortality, intraoperative and post-operative complications among the two study arms.
* To compare costs and cost-effectiveness between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Recurrent VC confirmed by histological examination
* Patient who underwent multiple treatments (surgery and radiation therapy or chemoradiation, radiation therapy or chemoradiation and chemotherapy).
* Patient not eligible for standard therapies (surgery, radiation therapy and systemic chemotherapy in case of metastatic disease) due to the performance status (ECOG Performance Status ≥ 3 )
* Life expectancy more than three months
* Measurable disease according to RECIST 1.1
* Adequate bone marrow, liver, and kidney function (creatinine <1.5 mg/dl), and coagulation parameters as follows:

  * Bone marrow (Hemoglobin ≥ 8.0 g/dL with or without transfusion support, Platelet count ≥ 75 × 109/L?) o INR >1.5;
  * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic-pyruvate transaminase (SGPT) ≤3.0 × upper limit of normal (ULN)
  * Total bilirubin ≤2.0 × ULN or ≤3 × ULN except for subjects with Gilbert's syndrome
  * Serum creatinine <1.5 mg/dl and creatinine clearance > 30 ml/min All blood assessments must be performed within 15 days from ECT treatment.
* For females of childbearing potential, a negative serum pregnancy human chorionic gonadotropin (hCG) pregnancy test within 72 hours of study Day 1.
* Signed informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply the study requirements.

Exclusion Criteria:

* History of other malignancies in the previous five years, except basal cell carcinoma of the skin.
* History of psychological, familial, sociological, or geographical condition potentially preventing compliance with the study protocol and follow-up schedule.
* Allergic reactions to the two chemotherapy drugs (BLM and AUC2-CARBOPLATIN) and/or their excipients.
* Evidence of pulmonary fibrosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Compare Local progression-free survival | 5 years
  Evaluate the oncology response to electroporation after administration of BLM + CBP to BLM alone in terms of local progression-free survival (LPFS) in women with relapsed vulvar cancer after multimodal treatments.

SECONDARY OUTCOMES:
Compare Health-Related Quality of life (HR-QoL) in patients undergoing BLM + AUC2-CARBOPLATIN vs BLM alone assessed with questionnaires in patients undergoing BLM + CBP vs BLM alone assessed with questionnaires. | 5 years
  Paper or electronic questionnaires will be given to the patient at baseline (within 30 days prior to randomization) and then at every follow-up visit within the first year after randomization.The significance and relevance of the data need to be explained carefully to participating patients so that they are motivated to comply with data collection. The patient must complete the questionnaire him/herself without receiving help from relatives, friends or clinic staff to answer the questionnaire. However, if the patient is unable to read the questionnaire (e.g., is blind or illiterate) the questionnaire may be read out by trained clinic staff and responses recorded.
Compare Health-Related Quality of life (HR-QoL) in the two study arms assessed with the EQ-5D-5L (5-level EQ-5D version) questionnaire. | 5 years
  The EQ-5D-5L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions.
Compare Health-Related Quality of life (HR-QoL) in the two study arms assessed with the FACT-V (Functional Assessment of Cancer Therapy-Vulva) questionnaire. | 5 years
  The FACT-V is a supplemental module that contains questions specifically related to the quality of life of patients with VC. The survey assesses the impacts of cancer therapy in four domains: physical, social/family, emotional, and functional. The response scale is a 5-point Likert type scale. The FACT-V is also has additional questions regarding issues that may be affected by vulvar cancer.
Compare Health-Related Quality of life (HR-QoL) in the two study arms assessed with the FACIT-PAL ( Functional Assessment of Chronic Illness Therapy - Palliative Care) questionnaire. | 5 years
  The FACIT-PAL ( is a 19-item palliative care subscale with items that pertain to persons with life-limiting illness. This questionnaire has items that pertain to symptoms that can be seen in advanced illness (e.g., shortness of breath, constipation, xerostomia), family and friend relationships (e.g., feeling appreciated by family, being a burden to family, maintaining contact with friends), life closure issues (e.g., having "made peace" with others, feeling hopeful, making "each day count"), and decision-making and communication abilities. The response scale is a 5-point Likert type scale.
Compare Overall Survival | 5 years
  To compare Overall Survival in the two study arms.
Reporting of Adverse Events and Serious Adverse Events | 5 years
  Toxicity will be evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events) criteria based on AE (Adverse Events) related or possibly related to the procedure and the drugs utilized, and to SAE (Serious Adverse Event) and AESI (Adverse Events of Special Interest), whether or not the event is considered treatment related.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS- Azienda Ospedaliera-Universitaria di Bologna, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: Undecided